CLINICAL TRIAL: NCT01490697
Title: Developing Memory Reconsolidation Blockers as Novel PTSD Treatments
Brief Title: Developing Memory Reconsolidation Blockers as Novel Posttraumatic Stress Disorder (PTSD) Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Roger K. Pitman, MD (Other)
Responsible Party: Sponsor-Investigator, Roger K. Pitman, MD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009P000647
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Post-traumatic Stress Disorder
Keywords: stress disorders; posttraumatic; memory; mifepristone; d-cycloserine; psychophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic | interventions — Mifepristone; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone plus d-Cycloserine (DCS) (Experimental): DCS 100 mg capsule orally followed by mifepristone1800 mg tablet orally 4 hours later and 90 minutes prior to traumatic memory retrieval via the traumatic event script preparation procedure, all on Day 7.
  Interventions: Drug: Mifepristone; Drug: d-Cycloserine
- Placebo plus Placebo (Placebo Comparator): Placebo-matching DCS 100 mg capsule orally followed by placebo-matching mifepristone1800 mg tablet orally 4 hours later and 90 minutes prior to traumatic memory retrieval via the traumatic event script preparation procedure, all on Day 7.
  Interventions: Drug: Placebo-matching Mifepristone; Drug: Placebo-matching d-Cycloserine (DCS)

INTERVENTIONS:
Drug: Mifepristone — 1800 mg tablet, single dose 90 minutes prior to script preparation on Day 7.
  Other Names: RU-486, Mifeprex
  Arms: Mifepristone plus d-Cycloserine (DCS)
Drug: d-Cycloserine — 100 mg capsule, single dose, taken 4 hours prior to to mifepristone on Day 7.
  Other Names: Seromycin
  Arms: Mifepristone plus d-Cycloserine (DCS)
Drug: Placebo-matching Mifepristone — Placebo-matching mifepristone tablets
  Arms: Placebo plus Placebo
Drug: Placebo-matching d-Cycloserine (DCS) — Placebo-matching DCS capsules
  Arms: Placebo plus Placebo

SUMMARY:
Despite substantial therapeutic advances, Posttraumatic Stress Disorder (PTSD) remains difficult to treat. One promising new area of research is in post-reactivation pharmacologic intervention, which is based upon the concept of blockade of memory reconsolidation. Recent animal research suggests that reactivation (retrieval) of a stored memory can return it to a labile (alterable) state from which it must be restabilized in order to persist. This process is called "reconsolidation," and various drugs have been found to block it in animals. This blockade may lead to a weakening of the original memory trace.

The aim of this study is to pilot the effect of mifepristone on physiologic responding during traumatic imagery. Although mifepristone is widely and safely used to cause a medical abortion, it is also a powerful stress hormone receptor blocker. These stress hormones, called glucocorticoids, may enhance memory (re)consolidation. Indeed, a recent study in animals reported that mifepristone blocked reconsolidation of context-conditioned fear in rats.

Reconsolidation blockade is a two-stage process. First, the memory must be destabilized by recalling it. Second, reconsolidation of the memory must be blocked by a drug. Memory traces formed under stressful conditions may resist destabilization and thus are inaccessible to reconsolidation blockers. However, when a reconsolidation blocker was paired with d-cycloserine (DCS) in animals that had been trained under stressful conditions, reconsolidation blockade became successful. These results suggest that DCS promotes the destabilization of resistant memory traces. The traumatic memories of individuals with PTSD may be particularly resistant to destabilization. Therefore, this study will compare mifepristone paired with DCS to placebo controls.

The same script-driven traumatic imagery method validated in previous studies of propranolol in this lab will be used. Briefly, subjects with PTSD will describe their traumatic event during a script preparation session, which will reactivate the memory. They will then receive a) mifepristone and DCS or b) placebo. A week later, they will engage in script-driven mental imagery of their traumatic event while physiologic responses (heart rate, sweating, etc) are measured. This is a pilot study so there are no formal hypotheses. The aim is to estimate effect sizes for mifepristone and to compare them with effect sizes for propranolol from this lab's previous work.

ELIGIBILITY:
Inclusion Criterion:

* Participant has experienced a traumatic event that meets the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV)11 A1. and A.2. PTSD criteria
* Participant currently meets DSM-IV criterion B.5, viz., "physiological reactivity on exposure to internal or external cues that symbolize or resemble an aspect of the traumatic event."

Exclusion Criteria:

* Medical condition that contraindicates the administration of mifepristone, e.g., history of adrenal failure; concurrent corticosteroid therapy; hemorrhagic disorders; cardiovascular, hypertensive, hepatic, respiratory or renal disease; insulin dependent diabetes mellitus; severe anemia; heavy smoking; porphyria; allergy to mifepristone; concurrent anticoagulant therapy; or medical condition that contraindicates the administration of DCS e.g., hypersensitivity to cycloserine, epilepsy, severe renal insufficiency.
* Pregnant (as determined by mandatory blood pregnancy testing, or currently breast feeding. (Note: Women who have had a hysterectomy or are post-menopausal (defined as over the age of 50 with no menstrual period for at least 12 months) will be exempted from pregnancy testing. Furthermore, women of childbearing potential will only be included if: a) they are using contraception in the form of barrier methods with spermicide, hormonal methods (e.g. birth control pill), or intrauterine devices (IUDs), or b) they have not been sexually active for the preceding 60 days.)
* Contraindicating psychiatric condition, e.g., current psychotic, bipolar, melancholic, or substance dependence or abuse disorder; or currently suicidal.
* Cognitive Impairment or dementia
* Initiation of, or change in, psychotropic medication within one month prior to recruitment
* Current use of medication that may involve potentially dangerous interactions with mifepristone, including certain CYP 3A4 substrates such as calcium channel blockers, azole antifungals, macrolide antibiotics, and tricyclic antidepressants. (Note - we have not included in this list benzodiazepines or selective serotonin reuptake inhibitors, because these drugs are frequently used by PTSD participants, and they have sufficiently wide therapeutic ranges such that any transient increases in blood levels induced by a single dose of mifepristone will not endanger participants); or current use of medication that may involve potentially dangerous interactions with DCS, including ethionamide, isoniazid, and pyridoxine.
* Inability to understand the study's procedures, risks, and side effects, or to otherwise give informed consent for participation;
* Age less than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Pitman, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dallas VA, Dallas, Texas

REFERENCES:
- [Result] Wood NE, Rosasco ML, Suris AM, Spring JD, Marin MF, Lasko NB, Goetz JM, Fischer AM, Orr SP, Pitman RK. Pharmacological blockade of memory reconsolidation in posttraumatic stress disorder: three negative psychophysiological studies. Psychiatry Res. 2015 Jan 30;225(1-2):31-39. doi: 10.1016/j.psychres.2014.09.005. Epub 2014 Sep 16. PMID 25441015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Plus Placebo | Mifepristone Plus d-Cycloserine (DCS)
Started | 16 | 18
Completed | 15 | 16
Not Completed | 1 | 2
Not completed — Did Not Meet PTSD Diagnostic Criteria | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants included in the analysis. 3 participants did not meet PTSD diagnostic criteria and are excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Placebo | Mifepristone Plus d-Cycloserine (DCS) | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (11.8) | 41.9 (13.9) | 38.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 7 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Physiological Posttraumatic Stress Disorder (PTSD) Probability as Determined From Psychophysiologic Responses to Traumatic Recollection
Description: The posterior probability of developing PTSD was determined for each participant from a composite of psychophysiological responses to script-driven imagery of traumatic events that included assessments of heart rate response in beats per minute, skin conductance response in microSiemens, and corrugator electromyogram (EMG) responses of the left lateral frontalis facial muscle in microVolts. Responses for the traumatic scripts were averaged and square-root transformed for analysis. Responses during personal traumatic imagery of previously studied individuals with and without current PTSD was used to calculate each participant's posterior probability of being classified as PTSD.
Time Frame: 1 week following treatment (Day 14)
Population: All randomized participants included in the analysis. Three participants did not meet PTSD diagnostic criteria and are excluded.
Measure: Mean (Standard Deviation); unit: percent probability
Arm/Group | Placebo Plus Placebo | Mifepristone Plus d-Cycloserine (DCS)
Number analyzed (Participants) | 15 | 16
percent probability | 44 (24) | 45 (22)
Statistical Analysis 1: Comparison: Placebo Plus Placebo vs Mifepristone Plus d-Cycloserine (DCS); Test type: Superiority; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-18 to 16] — Placebo plus Placebo - Mifepristone plus d-Cycloserine (DCS)

2. Secondary Outcome: Change From Baseline in the Impact of Event Scale-Revised (IES-R) Total Score
Description: IES-R is a 22-item patient reported measure of PTSD symptoms. Each question is answered using a 5-point scale where 0=not at all to 4=extremely for a total possible score of 0 to 88. Lower scores represent less severe symptoms and higher scores representing more severe symptoms. IES-R change scores were calculated by subtracting the Day 14 IES-R total score from the Day 7 IES-R total score. A negative change from Baseline indicates improvement of symptoms and a positive change from Baseline indicates a worsening of symptoms.
Time Frame: Day 7 (Baseline) and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Plus Placebo | Mifepristone Plus d-Cycloserine (DCS)
Number analyzed (Participants) | 15 | 16
score on a scale
  Baseline | 55.3 (21.9) | 52.4 (15.3)
  Change from Baseline at Day 14 | -5.0 (16.6) | -8.9 (11.9)
Statistical Analysis 1: Comparison: Placebo Plus Placebo vs Mifepristone Plus d-Cycloserine (DCS); Test type: Superiority; Mean Difference (Net) = 3.9, 95% CI 2-sided [-6.9 to 14.7] — Placebo plus Placebo - Mifepristone plus d-Cycloserine (DCS)

ADVERSE EVENTS:
Time Frame: 14 Days
Description: All randomized participants included in the analysis. Three participants did not meet PTSD diagnostic criteria and are excluded.
Arm/Group | Placebo Plus Placebo | Mifepristone Plus d-Cycloserine (DCS)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes